CLINICAL TRIAL: NCT03476707
Title: Association of Anemia With Hospital Costs in Elective Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM9
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Surgery; Surgical Blood Loss; Anemia; Colon Cancer; Economic Problems
MeSH Terms: conditions — Blood Loss, Surgical; Anemia; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anemic: People with a preoperative hematocrit less than 0.39
  Interventions: Other: Anemia
- Non-anemic: People with a preoperative hematocrit greater than or equal to 0.39

INTERVENTIONS:
Other: Anemia — Hematocrit less than 0.39
  Groups: Anemic

SUMMARY:
The objective is to measure the adjusted association between preoperative anemia and total hospital costs. We hypothesize that patients with anemia before surgery will have higher hospitalization costs than people without anemia.

DETAILED DESCRIPTION:
This study will examine the association between preoperative anemia (hematocrit less than 0.39; low blood counts) and hospital total costs from elective colorectal surgery. Total costs will be defined as the combination of direct and indirect costs ascertained using standardized patient-level costing algorithms (i.e. the standard way that hospital measure their costs). Adjustment will be made for factors that are likely to influence both the presence of anemia and costs of care.

ELIGIBILITY:
Inclusion Criteria:

* Elective hospital admission
* having colorectal surgery

Exclusion Criteria:

* not enrolled in national surgical quality improvement program data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults having elective colorectal surgery with national surgical quality improvement program data available
Sampling Method: Non-Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng S, Greenberg J, Moloo H, Thavorn K, McIsaac DI. Hospital cost associated with anemia in elective colorectal surgery: a historical cohort study. Can J Anaesth. 2019 Aug;66(8):877-885. doi: 10.1007/s12630-019-01379-8. Epub 2019 May 1. PMID 31044414

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anemic | Non-anemic
Started | 381 | 470
Completed | 381 | 470
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anemic | Non-anemic | Total
Number analyzed (Participants) | 381 | 470 | 851
Age, Customized [Count of Participants; unit: Participants]
  Age: < 65 | 123 | 272 | 395
  Age: 65-74 | 105 | 117 | 222
  Age: 75-84 | 114 | 67 | 181
  Age: >84 | 39 | 14 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 181 | 395
  Male | 167 | 289 | 456
Independent Functional Status [Count of Participants; unit: Participants] — Measure is based on NSQIP functional status definition (count of participants that are independent):
  Independent: The patient does not require assistance from another person for any activities of daily living. This includes a person who is able to function independently with prosthetics, equipment, or devices.
  Not independent: requires assistance for some or all activities of daily living
  Participants | 353 | 467 | 820
Elixhauser comorbidity index [Mean (Standard Deviation); unit: Index] — The Elixhauser Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases diagnosis codes. Each comorbidity category is documented as disease presence or disease absence and there are 31 categories. Therefore, a higher score indicates more presence of disease (worse outcome) (with 31 being the maximum and 0 being the minimum).
  Index | 6.16 (5.98) | 5.50 (5.89) | 6 (6)
Procedural Index for Mortality Risk (PIMR) Score [Mean (Standard Deviation); unit: Number of procedural risk points] — An index that quantifies the relative contribution of a broad range of therapeutic procedures on the risk of death in hospital. Score values range from -7 to +11 (higher score indicates greater risk).
  Number of procedural risk points | 0.47 (1.39) | 0.17 (0.70) | 0.3 (1.1)
American Society of Anesthesiology (ASA) Score [Count of Participants; unit: Participants] — Physical status classification used to determine a patient's risk with anaesthesia. The score ranges from I to VI, with I indicating a healthy person and VI indicating a deceased organ donor. A higher score indicates greater risk.
  Participants
    I-II | 51 | 142 | 193
    III | 260 | 302 | 562
    IV-V | 70 | 26 | 96

OUTCOME MEASURES:

1. Primary Outcome: Total Hospital Costs
Description: Direct and indirect costs accrued during the index hospitalization. Costs were measured using standard and validated algorithms, standardized to 2016 CAD. This method accounts for a patient's resource intensity weight, their case mix group, as well as fixed patient costs (e.g., medications, investigations) and indirect costs to the hospital based on patient's location of care (intensive care unit versus ward) and length of stay.
Time Frame: Hospital admission to date of discharge from hospital, or 365 days after admission, whichever came first
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Anemic | Non-anemic
Number analyzed (Participants) | 381 | 470
Dollars | 23,667 (32,210) | 17,100 (10,822)

2. Secondary Outcome: Length of Stay
Description: Number of days in hospital after surgery
Time Frame: Date of surgery to date of hospital discharge, or up to one year after surgery (whichever comes first)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Anemic | Non-anemic
Number analyzed (Participants) | 381 | 470
Days | 12.4 (17.5) | 8.5 (7.5)

3. Secondary Outcome: Red Blood Cell Transfusion
Description: Any red blood cell transfusion received
Time Frame: Hospital admission to date of surgery, or 365 days after admission, whichever came first
Measure: Count of Participants; unit: Participants
Arm/Group | Anemic | Non-anemic
Number analyzed (Participants) | 381 | 470
Participants | 88 | 18

ADVERSE EVENTS:
Time Frame: AEs were not collected
Description: AEs were not expected or collected.
Arm/Group | Anemic | Non-anemic
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Findings may not be generalizable to other jurisdictions with different hospital funding models and findings provide only an association between anemia and costs. There is risk of confounding bias due to unmeasured variables that might influence the presence of anemia or the accumulation of costs. The lack of integration of transfusion costs in our healthcare system required us to estimate the added cost of transfusions, and we were also unable to account for physician remuneration costs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No